CLINICAL TRIAL: NCT00461604
Title: High Dosage Esomeprazole and Baclofen for Therapy of Gastroesophageal Reflux Disease
Acronym: NEXBAC
Status: Completed | Type: Observational
Sponsor: Technical University of Munich (Other)
Responsible Party: Technische Universität München, II. Medizinische Klinik, Technische Universität München
Other Study IDs: 1690/07
Record Dates: First submitted 2007-04-16; First posted 2007-04-18 (Estimated); Last update posted 2008-05-20 (Estimated); Status verified 2008-05

CONDITIONS: Patients With Persistent Objectified Gastroesophageal Reflux and Reflux-Associated Symptoms Despite PPI-Therapy With 40mg Esomeprazole
Keywords: gastroesophageal reflux disease; baclofen; impedance
MeSH Terms: conditions — Gastroesophageal Reflux

STUDY DESIGN:
Time Perspective: Prospective
Oversight: Data Monitoring Committee: Yes

SUMMARY:
It has been reported that Baclofen is an appropriate tool in the therapeutic management of Gastroesophageal Reflux Disease. To objectify gastroesophageal reflux combined pH-metry/impedance monitoring was applied to patients with persistent reflux-associated symptoms despite PPI-therapy (40mg esomeprazole for 2 weeks). After provement of pathological findings in the test PPI-dosage was escalated to double standard-dosage for another for weeks. In case of persistent symptoms another ph-metry/impedance monitoring was performed. In case of pathological findings additional baclofen was administered to the therapeutic regime. After 3 months another ph-metry/impedance monitoring was performed. At the time point of the tests a questionnaire was completed.

Aim of the study was to evaluate the influence of high dosage PPI-therapy and additional baclofen in patients with persistent symptoms and objectified gastroesophageal reflux.

ELIGIBILITY:
Inclusion Criteria:

* age between 18-70 years
* informed consent
* patients with persistent reflux-associated symptoms despite PPI-therapy

Exclusion Criteria:

* epilepsy
* synthetic liver diseases
* renal failure
* disability to understand informed consent

Ages: 18 Years to 70 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 40 (Estimated)
Dates: Start 2006-10; Primary Completion 2008-05 (Actual); Study Completion 2008-05 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Alexander Meining, MD, Principal Investigator — Technische University Munich
Locations (1):
- Technical University of Munich, Munich, Bavaria, Germany